CLINICAL TRIAL: NCT03194126
Title: Evaluation of Efficacy of Two Therapeutic Strategies for Cervical Maturation Before Medical Termination: Mechanical Plus Medicinal Maturation vs Medicinal Maturation Alone
Brief Title: Evaluation of Efficacy of Two Therapeutic Strategies for Cervical Maturation Before Medical Termination
Acronym: IMEGYN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LOCAL/2016/VL-01
Record Dates: First submitted 2017-06-16; First posted 2017-06-21 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Medical; Abortion, Fetus
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary outcome will be evaluated by a blinded evaluator: the laminaria placement is performed by the on-call team at Day-1, whilst the delivery is performed by a different team at Day 0, with the laminaria removed in the morning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mifepristone + Misoprostol OR oxytocine + laminaria (Experimental)
  Interventions: Procedure: Mifepristone + Misoprostol OR oxytocine + laminaria
- Mifepristone + Misoprostol OR oxytocine (Other)
  Interventions: Procedure: Mifepristone + Misoprostol OR oxytocine

INTERVENTIONS:
Procedure: Mifepristone + Misoprostol OR oxytocine + laminaria — Three laminaria placed 12 hours prior to administration of misoprostol
  Arms: Mifepristone + Misoprostol OR oxytocine + laminaria
Procedure: Mifepristone + Misoprostol OR oxytocine — standart support
  Arms: Mifepristone + Misoprostol OR oxytocine

SUMMARY:
Reducing the time patients spend in the labor and delivery room saves money and reduces patient discomfort as well and reducing complications. We will compare two methods for inducing cervical maturation in order to shorten the time taken between administration of drugs and delivery.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patients is at least 18 years old
* Patient with a singleton pregnancy between 14 and 34 weeks gestation with an indication for medical termination due to maternal or fetal problem as validated by pluridisciplinary prenatal diagnosis center.

Exclusion Criteria:

* The subject is participating in an interventional study or is in a period of exclusion determined by a previous study
* The patient is under safeguard of justice
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* Patient has vaginismus
* Patient has a cervix permitting artificial rupture of membrane
* Patients taking one of the following treatments, contraindicated for mifepristone: ketoconazole, itraconazole, erythromycin, grapefruit juice, rifampicin, dexamethasone, St John's wort and certain anti-convulsants (phenytoin, phenobarbital, carbamazepine).

Patients contraindicated for oxytocine.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-02-11 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
time taken between administration of 1st dose of drugs and delivery between the two strategies | Up to 2 days

SECONDARY OUTCOMES:
Compare pain experienced by patients between groups | Day 0 - Day 2
  scale 0-10
Compare cervix length before administration of Misoprostol OR oxytocine between groups | Day 0
  in mm
Compare degree of dilation before administration of Misoprostol OR oxytocine between groups | Day 0
  in cm
Compare time taken between Misoprostol OR oxytocine and delivery between groups | Day 0 - Day 2
  hours
Rate of delivery between groups | 4 hours
Rate of delivery between groups | 6 hours
Rate of delivery between groups | 8 hours
Rate of delivery between groups | 12 hours
Rate of delivery between groups | >12 hours
Incidence of endometritis between groups | Day 0 - Day 2
Incidence of hemorrhage between groups | Day 0 - Day 2
Patient satisfaction in peripartum between groups | Day 2
  Numeric Rating Scale (0-10)
Patient anxiety between groups | Day 0 - 3 months
  Hospital Anxiety and Depression Scale questionnaire
Evaluation of any post-traumatic stress between groups | 3 months
  Perinatal post-traumatic stress disorder questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Montpellier, Montpellier
  - CHU Nimes, Nîmes

IPD SHARING:
Plan to Share IPD: No